CLINICAL TRIAL: NCT00003721
Title: A Phase I, Pharmacologic and Biologic Study of Col-3 (NSC683551) Administered on a 28-Day Oral Dosing Schedule in Patients With Advanced Solid Tumors
Brief Title: Chemotherapy in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066830; U01CA069853 (NIH); P30CA054174 (NIH); UTHSC-9785011153 (Other: UTHSCSA IRB); SACI-IDD-97-27 (Other: San Antonio Cancer Institute); NCI-T97-0091 (Other: NCI)
Record Dates: First submitted 1999-11-01; First posted 2004-02-09 (Estimated); Last update posted 2012-06-29 (Estimated); Status verified 2012-06

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: incyclinide — This is a dose escalation study. Patients receive oral COL-3 once daily. Treatment continues in the absence of disease progression and unacceptable toxic effects. Cohorts of 3-6 patients each receive escalating doses of COL-3. Dose escalation to the next level occurs after 3 patients have completed 28 days of treatment without dose limiting toxicity (DLT). Dose escalation continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience DLT.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of COL-3 in treating patients who have advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES: I. Define the maximum tolerated dose of COL-3 in patients with advanced solid tumors. II. Identify the dose limiting toxicity and safety profile of COL-3 in these patients. III. Define the pharmacokinetics and pharmacodynamics of COL-3 in these patients. IV. Observe any evidence of antitumor activity through standard response criteria or biologic surrogate markers.

OUTLINE: This is a dose escalation study. Patients receive oral COL-3 once daily. Treatment continues in the absence of disease progression and unacceptable toxic effects. Cohorts of 3-6 patients each receive escalating doses of COL-3. Dose escalation to the next level occurs after 3 patients have completed 28 days of treatment without dose limiting toxicity (DLT). Dose escalation continues until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 or more of 6 patients experience DLT.

PROJECTED ACCRUAL: Up to 30 patients will be accrued within 1 year for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically or cytopathologically proven advanced solid tumors for which no conventional therapy exists or that is refractory to standard therapy No primary brain tumors or active brain metastases, including known evidence of cerebral edema by CT or MRI, known tumor progression from prior imaging studies or clinical symptoms of/from brain metastases

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0-2 Life expectancy: Greater than 12 weeks Hematopoietic: Absolute neutrophil count greater than 1,500/mm3 Platelet count greater than 100,000/mm3 Hemoglobin greater than 9 g/dL Hepatic: Bilirubin normal PT or PTT normal ALT or AST less than 2.5 times upper limit of normal Renal: Creatinine less than 1.5 mg/dL OR Creatinine clearance greater than 60 mL/min Cardiovascular: No myocardial infarction, stroke, or congestive heart failure within 3 months Other: HIV negative Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No history of gastrointestinal disorders that interfere with absorption of COL-3 No active infections or other medical illnesses No psychological or social problems No emotional disorder or substance abuse No hypersensitivity to tetracycline or its derivative

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since chemotherapy At least 6 weeks since nitrosoureas or mitomycin At least 3 months since suramin Endocrine therapy: No concurrent steroids Radiotherapy: At least 4 weeks since prior large field radiation therapy (greater than 20% of total bone marrow) Surgery: At least 14 days since major surgery No major upper gastrointestinal surgery Other: No concurrent anticonvulsant medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 1998-11; Primary Completion 2002-04 (Actual); Study Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric K. Rowinsky, MD, Study Chair — San Antonio Cancer Institute
Locations (1):
- San Antonio Cancer Institute, San Antonio, Texas, United States